CLINICAL TRIAL: NCT06202430
Title: Comparison of Ultrasound Guided High Thoracic Erector Spinae Plane Block With Shoulder Block for Postoperative Analgesia in Arthroscopic Shoulder Surgery
Brief Title: Ultrasound Guided Block for Postoperative Analgesia in Arthroscopic Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Nevine Mostafa Soliman, Lecturer of Anesthesiology, ICU and Pain Management., Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122023ANET14
Record Dates: First submitted 2023-12-27; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided High Thoracic Erector Spinae Plane Block (Active Comparator): High Thoracic-ESPB The patient was placed in the lateral decubitus. Subsequently, an ultrasound (US)-guided aseptic technique, with a high-frequency linear probe enveloped in a sterile sheath containing a thin film of US gel, was used to locate the transverse process of T2. After LA skin infiltration, a 22-G block was inserted in a cephalocaudal direction until the space between the fascia of the erector spinae and the transverse process of T2 was identified. After negative aspiration, hydro dissection using 2 mL of saline was performed. Eventually, 30 mL of the LA bupivacaine 0.25% and epinephrine 5 µg/ mL was injected.
  Interventions: Procedure: High Thoracic Erector Spinae Plane Block
- Ultrasound Guided Shoulder Block (Active Comparator): Shoulder Block Suprascapular nerve block (SSNB) approach: A high-frequency linear probe was utilized across the supra-spinous fossa parallel to the spine of the scapula after skin cleaning with an antiseptic solution, if a deep block is required, a low frequency probe was required. A hyperechoic line was identified, followed by an acoustic shadow that corresponds to the floor of the supra-spinous fossa. The needle was progressed in plane from medial to lateral after local infiltration of the skin with 1% lidocaine. We directed the needle towards the lateral side of the supra-spinous fossa if the neuro-vascular bundle was not evident. After careful aspiration, 10 ml of 0.5% bupivacaine was injected under the supraspinatus muscle. Along with Axillary nerve block technique.
  Interventions: Procedure: Shoulder Block

INTERVENTIONS:
Procedure: High Thoracic Erector Spinae Plane Block — High Thoracic-ESPB The patient was placed in the lateral decubitus. The transverse process of T2 was identified. After negative aspiration, hydro dissection using 2 mL of saline was performed. Eventually, 30 mL of the LA bupivacaine 0.25% and epinephrine 5 µg/ mL was injected.
  Arms: Ultrasound Guided High Thoracic Erector Spinae Plane Block
Procedure: Shoulder Block — Shoulder Block Suprascapular nerve block (SSNB) approach: The needle was progressed in plane from medial to lateral after local infiltration of the skin with 1% lidocaine. We directed the needle towards the lateral side of the supra-spinous fossa if the neuro-vascular bundle was not evident. After careful aspiration, 10 ml of 0.5% bupivacaine was injected under the supraspinatus muscle.
  Axillary nerve block technique:
  The nerve approach had been described in plane from cranial to caudal. After local infiltration of the skin with 1% lidocaine, the needle tip must be visualized within the fascia below the teres minor muscle and just above the PCHA. After cautious aspiration, 10 ml of 0.5% bupivacaine was injected on the posterior aspect of the humerus.
  Arms: Ultrasound Guided Shoulder Block

SUMMARY:
This study aimed to compare the efficacy of high thoracic-ESPB with shoulder block as analgesic options for arthroscopic shoulder surgery.

Primary outcome:

• 24-hour analgesic consumption.

Secondary outcomes:

* Postoperative pain evaluated by: Visual Analogue Pain Scale (VAS).
* Time to first rescue analgesia and total postoperative consumption of analgesia.
* Effect of the block on Hemodynamics.
* Adverse effects in the form of postoperative nausea and vomiting (PONV).
* Patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All patients within the age range ≥ 21 to ≤ 70 years old.
* Body mass index (BMI) ≤ 35kg m2.
* ASA I, II of both sex

Exclusion Criteria:

* Refusal of the patient to the study.
* Infection at the site of injection.
* Previous known allergy to any drug used in the study by history.
* Renal disease [Creatinine. >3mg/dl.].
* Hepatic disease. [ALT>50U/L, AST >50U/L].
* Un cooperative or psychological unstable patients.
* Coagulopathy or anticoagulant therapy.
* Pregnancy.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-13 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
24-hour analgesic consumption. | 24 hours.
  Total consumptive dose of Morphine. Patients started acetaminophen (1 g PO) before surgery. Acetaminophen infusion continued postoperatively at a dose of 1 g/6 hours. Later, 75 mg diclofenac sodium was also given intravenously twice a day, in combination with 40 mg pantoprazole once. Rescue analgesia of 2.5 mg morphine was given intravenously if the postoperative Visual Analogue Scale score was > 3 or the patient requested additional analgesia.

SECONDARY OUTCOMES:
Visual Analogue Scale. | ● Every 0.5 hour for next 2 hours. ● Every 2 hours for next 6 hours. ● Every 6 hours for remaining 24 hours post-operatively.
  The pain control target was considered at Visual Analogue Scale score (VAS) < 4, where VAS score of 0 means no pain and VAS score of 10 means the worst pain imaginable. Postoperative pain evaluated by: Visual Analogue Pain Scale (VAS).
  Time to first rescue analgesia and total postoperative consumption of analgesia.
  Effect of the block on Hemodynamics. Adverse effects in the form of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- MenoufiaU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided